CLINICAL TRIAL: NCT05447364
Title: Efficacy of Different Doses of Pregabalin as a Multimodal Analgesic Agent in Postoperative Pain Control After Total Knee Arthroplasty - A Randomized Controlled Trial
Brief Title: Efficacy of Different Doses of Pregabalin as a Multimodal Analgesic Agent in Postoperative Pain Control After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Seksan Kukreja, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-OT-6-150/64
Record Dates: First submitted 2022-06-26; First posted 2022-07-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Pregabalin
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Participants are randomized and assigned to 75 mg of Pregabalin and 150 of Pregabalin groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 75 mg of Pregabalin (Experimental): Participant received 1 tab of 75 mg of Pregabalin and 1 tab of placebo
  Interventions: Drug: Pregabalin 75mg
- 150 mg of Pregabalin (Active Comparator): Participant received 2 tabs of 75 mg of Pregabalin
  Interventions: Drug: Pregabalin 150mg

INTERVENTIONS:
Drug: Pregabalin 75mg — 1 tab of Pregabalin Brillior 75 mg and 1 tab of Placebo
  Arms: 75 mg of Pregabalin
Drug: Pregabalin 150mg — 2 tabs of Pregabalin Brillior 75 mg
  Arms: 150 mg of Pregabalin

SUMMARY:
The purpose of this study is to compare the efficacy of 75 mg of Pregabalin and 150 mg of Pregabalin in postoperative pain control after TKA.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be chosen for eligibility for the study entry. At the day before surgery date, patients who meet the eligibility criteria will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to 75 mg of Pregabalin and 150 mg of Pregabalin groups.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic primary knee osteoarthritis undergoing unilateral TKA
2. Aged between 55 and 80 years old
3. Comply with protocol

Exclusion Criteria:

1. Allergy to any of the medications in this protocol (Pregabalin, Morphine, Paracetamol, Celecoxib, Tramadol, Aspirin)
2. Secondary osteoarthritis of the knee including autoimmune diseases and post-traumatic
3. Previous surgery on the knee
4. Contraindicated to spinal anesthesia (SB) or Adductor canal block (ACB)
5. GFR < 30ml/min, Severe Liver Function (Child-Pugh C)
6. History of seizure or cerebrovascular diseases

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Difference on 100-mm Visual analog scale (VAS) Pain Score between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 6, 12, 18, 24, 48 hours & 2, 6, 12 weeks after surgery
  * The 100-mm VAS pain score is a self-reported instrument assessing pain scores.
  * Participants will assess the VAS pain score at rest and on-movement
  * VAS Pain at rest is evaluated when the participant is at rest.
  * VAS Pain on-movement is evaluated on active extension and flexion of the operated knee using mean scores between the two.
  * Possible scores range from 0 (no pain) to 100 (worst imaginable pain)
  * Higher scores mean a worse pain

SECONDARY OUTCOMES:
Difference on Morphine consumption between 75 mg of Pregabalin and 150 mg of Pregabalin groups | From postoperative period until 48 hours after surgery
  Amount of Morphine consumption as rescue pain control reported as mg per day
Difference on side effects between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 6, 12, 18, 24, 48 hours & 2, 6, 12 weeks after surgery
  Common of side effects of Pregabalin and Morphine including sedation, dizziness, visual disturbances, nausea and vomiting
Difference on length of stay between 75 mg of Pregabalin and 150 mg of Pregabalin groups | From postoperative period until 48 hours after surgery
  Time to discharge
Difference on time to ambulation between 75 mg of Pregabalin and 150 mg of Pregabalin groups | From postoperative period until 48 hours after surgery
  Time from operation to ambulation before hospital discharge
Difference on Range of motion between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 2, 6, 12 weeks after surgery
  - Flexion and extension angle of the knee is measured by a long-arm goniometer
Difference on Knee Society Score between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 2, 6, 12 weeks after surgery
  * The Knee Society Score is a validated, objective scoring system to evaluate patient's functional abilities before and after total knee arthroplasty
  * The Knee Society Score has 2 sections including Knee Score and Functional Score with both sections scored from 0 to 100
  * Higher scores on the Knee Society Score indicate better knee conditions
Difference on Knee injury and Osteoarthritis Outcome Score between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 2, 6, 12 weeks after surgery
  * The Knee injury and Osteoarthritis Outcome Score is a validated, patient reported joint-specific score to assess patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items)
  * The Knee injury and Osteoarthritis Outcome Score range from 0 to 100
  * Higher scores on the Knee injury and Osteoarthritis Outcome Score indicate better knee conditions
Difference on Time up-and-go test between between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 2, 6, 12 weeks after surgery
  * The Time up-and-go test (TUGT) measures the time (seconds) that the patient takes to rise from a chair and walk for 3 meters. Then, he or she turns around and comes back to the seat at the initial position.
  * They were permitted to use walking aids if they wished.
  * TUGT was a reliable and valid test for quantifying functional mobility.
Difference on 2-minutes walking test between 75 mg of Pregabalin and 150 mg of Pregabalin groups | 2, 6, 12 weeks after surgery
  * Participants were instructed to walk for 2 minutes at their normal pace up and down a designated corridor, turning around at each end of the corridor without stopping
  * They were permitted to use walking aids if they wished.
  * The results were recorded as the total distance walked in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University Hospital, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: * Researchers who provide a methodologically sound proposal.
  * To achieve aims in the approved proposal.
  * Proposals should be directed to thesekku@gmail.com.
  * To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Mishriky BM, Waldron NH, Habib AS. Impact of pregabalin on acute and persistent postoperative pain: a systematic review and meta-analysis. Br J Anaesth. 2015 Jan;114(1):10-31. doi: 10.1093/bja/aeu293. Epub 2014 Sep 10. PMID 25209095
- [Result] Golladay GJ, Balch KR, Dalury DF, Satpathy J, Jiranek WA. Oral Multimodal Analgesia for Total Joint Arthroplasty. J Arthroplasty. 2017 Sep;32(9S):S69-S73. doi: 10.1016/j.arth.2017.05.002. Epub 2017 May 11. PMID 28705543
- [Result] Schmidt PC, Ruchelli G, Mackey SC, Carroll IR. Perioperative gabapentinoids: choice of agent, dose, timing, and effects on chronic postsurgical pain. Anesthesiology. 2013 Nov;119(5):1215-21. doi: 10.1097/ALN.0b013e3182a9a896. No abstract available. PMID 24051389
- [Result] Summers S, Mohile N, McNamara C, Osman B, Gebhard R, Hernandez VH. Analgesia in Total Knee Arthroplasty: Current Pain Control Modalities and Outcomes. J Bone Joint Surg Am. 2020 Apr 15;102(8):719-727. doi: 10.2106/JBJS.19.01035. No abstract available. PMID 31985507
- [Result] Buvanendran A, Kroin JS, Della Valle CJ, Kari M, Moric M, Tuman KJ. Perioperative oral pregabalin reduces chronic pain after total knee arthroplasty: a prospective, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):199-207. doi: 10.1213/ANE.0b013e3181c4273a. Epub 2009 Nov 12. PMID 19910619
- [Result] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Result] Jain P, Jolly A, Bholla V, Adatia S, Sood J. Evaluation of efficacy of oral pregabalin in reducing postoperative pain in patients undergoing total knee arthroplasty. Indian J Orthop. 2012 Nov;46(6):646-52. doi: 10.4103/0019-5413.104196. PMID 23325966
- [Result] Azboy I, Groff H, Goswami K, Vahedian M, Parvizi J. Low-Dose Aspirin Is Adequate for Venous Thromboembolism Prevention Following Total Joint Arthroplasty: A Systematic Review. J Arthroplasty. 2020 Mar;35(3):886-892. doi: 10.1016/j.arth.2019.09.043. Epub 2019 Oct 5. PMID 31733981
- [Result] Noiseux NO, Callaghan JJ, Clark CR, Zimmerman MB, Sluka KA, Rakel BA. Preoperative predictors of pain following total knee arthroplasty. J Arthroplasty. 2014 Jul;29(7):1383-7. doi: 10.1016/j.arth.2014.01.034. Epub 2014 Feb 7. PMID 24630598
- [Result] Unnanuntana A, Ruangsomboon P, Keesukpunt W. Validity and Responsiveness of the Two-Minute Walk Test for Measuring Functional Recovery After Total Knee Arthroplasty. J Arthroplasty. 2018 Jun;33(6):1737-1744. doi: 10.1016/j.arth.2018.01.015. Epub 2018 Jan 31. PMID 29454556
- [Result] YaDeau JT, Lin Y, Mayman DJ, Goytizolo EA, Alexiades MM, Padgett DE, Kahn RL, Jules-Elysee KM, Ranawat AS, Bhagat DD, Fields KG, Goon AK, Curren J, Westrich GH. Pregabalin and pain after total knee arthroplasty: a double-blind, randomized, placebo-controlled, multidose trial. Br J Anaesth. 2015 Aug;115(2):285-93. doi: 10.1093/bja/aev217. PMID 26170351